CLINICAL TRIAL: NCT03233763
Title: Laboratory Studies Into the Pathology of Leukaemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR4508
Record Dates: First submitted 2017-01-18; First posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bone Marrow and blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Bone Marrow Aspirate — Diagnostic Bone Marrow aspirate

SUMMARY:
Ongoing laboratory work into the pathology of Leukaemia:

DETAILED DESCRIPTION:
The investigators will test AML samples sent to the diagnostic laboratory from participants with newly diagnosed or relapsed/refractory AML. Samples will be sent from district general hospitals and teaching hospitals.

Results will be returned to referring clinicians in the same way investigators currently return results for samples sent for standard tests. The service will be advertised through the Royal Marsden Website with visibility to both participants and HCPs). The investigators will also inform all the clinicians involved in the AML working party (Dr Taussig is a member of the AML working group).

In addition we are looking at diagnostic approaches to IDH 1 and 2 mutation identification.

An initial comparison of 50 samples by three analysis methods will be conducted.

IDH1 and IDH2 variant discovery will first be performed using an established standard in house SOP (SOP: SMD103) for CE-SSCA

ELIGIBILITY:
Inclusion Criteria:

18 & Over Diagnosis of AML Generic Research consent given

Exclusion Criteria:

Under 18 No generic research consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an exploratory laboratory study using stored tissue where consent has already been given.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-04-24 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Pathology of Leukaemia cells | 15 years
  Pathology of Leukaemia cells

CONTACTS AND LOCATIONS:
Overall Officials: David Taussig, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Department of Haematology, the Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to patient tissue is via formal request to the Sponsor